CLINICAL TRIAL: NCT01899131
Title: A Prospective Clinical and Radiographic Assessment on New Platform-switched Laser Lok Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC 13 AS 177-13-TLV CTIL
Record Dates: First submitted 2013-06-26; First posted 2013-07-15 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2013-06

CONDITIONS: Preserve Crestal Bone Level and Gingival Margin Around Dental Implants
Keywords: dental implants; crestal bone; gingival margin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- platform-switch tapered internal implants (Other): 2 platform-switch tapered internal implants placed in 10 participants.clinical and radiographic assessment in 6,12,24, month post implant insertion
  Interventions: Device: platform-switch tapered internal implants

INTERVENTIONS:
Device: platform-switch tapered internal implants — Laser-Lok permanent abutment/ new Laser Lok platform-switch implant assembly.assessment at 6,12,24 month clinicaly and radiographic
  Other Names: Biohorizons platform-switch tapered internal implants

SUMMARY:
1. To investigate the hard and soft tissue adaptation and maintenance to the Laser-Lok® microchannels permanent abutment/ new Laser-Lok® implant assembly by performing clinical and radiographic evaluations.
2. To investigate the effect of inter-implant spacing (minimum of 2 or 3 mm) on hard and soft tissues.
3. To perform clinical and radiographic evaluations on these abutment/implant assemblies up to 2 years.

DETAILED DESCRIPTION:
* Screening (Inclusion/ Exclusion Criteria)
* Day of Surgery: Dental CT scan/ periapical radiograph / clinical picture / clinical examination (probing depth, BOP, gingival recession).
* Implant Restoration Day: Post-restoration periapical radiograph/ clinical picture/ clinical examination (probing depth, BOP, gingival recession).
* 6 month, 1 Year and 2 Year Post Restoration: periapical radiograph / clinical picture / clinical examination (probing depth, BOP, gingival recession).

ELIGIBILITY:
Inclusion Criteria:1. Male or female, between 20-70 years of age, who request dental implant treatment options for rehabilitation.

2. Subjects who are willing to sign an informed consent, participate and return for follow-up visits.

3. Subjects without significant medical history and currently not on medications that might complicate the results.

4. Subjects presenting with an edentulous area requiring a tooth-replacement option.

-

Exclusion Criteria:1. Subjects who do not meet all the inclusion criteria or who will not cooperate with the protocol schedule.

2. Subjects who received and failed a previously placed dental implant. 3. Subjects who require an onlay ridge augmentation procedure in the area to achieve adequate bone volume for the placement of dental implants.

4. Subjects who have significant untreated periodontal disease, caries, infection or chronic inflammation in the oral cavity within two adjacent tooth positions of the clinical trial area.

5. Subjects who have used nicotine-containing products within 3 weeks prior to surgery.

6. Subjects who are insulin-dependent diabetic or if their Hgb1c levels > 6.5%. 7. Subjects who have had a history of malignancy within the past 5 years (except for basal or squamous cell carcinoma of the skin or in situ cervical carcinoma).

8. Subjects who are nursing or pregnant. 9. Subjects who are presently taking medications (except estrogen/progesterone therapy) or those who are undergoing treatment that in known to have an effect on bone turnover.

10. Subjects who have diseases that affect bone metabolism (excluding idiopathic osteoporosis).

11. Subjects with a history of an autoimmune disease, documented allergy or multiple allergies to any component of the agents used in this study.

12. Acutely infected defect site. 13. Immediate implant site.

-

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
epithelial attachment and bone level around implants | 2 years
  prevent apical migration of the epithelial attachment, and preserve bone level around implant head. radiographic and clinical assessment during recall periods

SECONDARY OUTCOMES:
inhibit the loss of crestal bone . | 2 years
  preserve the coronal level of bone

CONTACTS AND LOCATIONS:
Overall Officials: Amnon Singer, DMD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel